CLINICAL TRIAL: NCT05093842
Title: Sedentary Behavior Reduction in Pregnancy Intervention Study
Acronym: SPRING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Bethany Barone Gibbs, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY20110193; AHA 20TPA35490099 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2021-09-23; First posted 2021-10-26 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-12

CONDITIONS: Pregnancy Complications; Sedentary Behavior
Keywords: Behavioral Intervention; Randomized Clinical Trial; Pregnancy
MeSH Terms: conditions — Pregnancy Complications; Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research personnel conducting outcome assessments will be blinded to participant group assignment. As the participant will be receiving a behavioral intervention, both the participant and interventionist will be aware of group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sedentary Behavior Reduction Intervention (Experimental): Biweekly virtual health coaching, height-adjustable work station, and fitbit - targetting decreasing sedentary behavior, increasing standing, and increasing steps per day. Printable information on physical activity recommendations also provided.
  Interventions: Behavioral: Sedentary Behavior Reduction; Behavioral: Information on Physical Activity Recommendations during Pregnancy
- Usual Care Control (Active Comparator): Printable information on physical activity recommendations only
  Interventions: Behavioral: Information on Physical Activity Recommendations during Pregnancy

INTERVENTIONS:
Behavioral: Sedentary Behavior Reduction — Participants receive bimonthly behavioral health coaching, a sit-stand desk attachment or table, and an activity prompter if they do not already have one (e.g., fitbit, as needed).
  Arms: Sedentary Behavior Reduction Intervention
Behavioral: Information on Physical Activity Recommendations during Pregnancy — Participants in the study will receive educational materials provided one time by email about the currently recommended physical activity during pregnancy.

SUMMARY:
This pilot and feasibility study will enroll newly pregnant women at risk for high sedentary behavior (SED) and elevated APO risk (n=53) and will randomize them to either a SED reduction intervention or control. Research aims include to: 1) demonstrate our ability to decrease SED and increase standing and light activity in pregnant women; 2) evaluate feasibility; and 3) gather preliminary effects on clinical outcomes including APOs, cardiometabolic risk factors, well-being, and fetal outcomes.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) accounts for 1 in 4 deaths among women of reproductive age. Decreasing adverse pregnancy outcomes (APO), e.g. hypertensive disorders of pregnancy, gestational diabetes, and preterm birth, could reduce this burden. APOs have serious immediate health consequences and are recognized by the AHA as major risk factors for future CVD. Yet, APOs are hard to prevent and treat, with a 20% prevalence that is increasing in the U.S. Moderate-vigorous intensity physical activity (MVPA) reduces APOs, but less than 1 in 4 pregnant women achieve guidelines and pregnant women report unique barriers such as fatigue, pain, medical restriction, and concern for the baby.

Sitting, or 'sedentary behavior' (SED) is a novel risk factor for CVD. Yet, sparse research and no U.S. guidelines exist for SED in pregnancy. Our recent AHA-funded cohort study in pregnant women (n=120) objectively measured SED and MVPA during each trimester. While MVPA was not related to outcomes, pregnant women with high vs. low SED across pregnancy had greater odds of APO and gave birth to babies at a reduced gestational age. Considering that decreasing SED may be more feasible given the barriers to MVPA, the investigators hypothesize that a SED reduction intervention may be especially promising for reducing APOs and improving cardiovascular health for women and their children.

Given the dearth of SED research, trials, or guidelines for pregnant women, the investigators propose to use our preliminary data on behavioral targets, correlates, and determinants of SED during pregnancy to adapt our previously successful SED reduction interventions. This pilot and feasibility study will enroll newly pregnant women with high SED and elevated APO risk (n=53) and randomize them to either a SED reduction intervention or control (2:1 ratio). Research aims include to: 1) demonstrate our ability to decrease SED and increase standing and light activity in pregnant women; 2) evaluate feasibility; and 3) gather preliminary effects on clinical outcomes including APOs, cardiometabolic risk factors, well-being, and fetal outcomes.

Participants will complete three assessment visits, one in each trimester, including 1-week monitoring of SED and activity patterns with a thigh-worn activPAL and blood pressure measurement using a standard protocol. Other outcomes will be assessed by self-report and medical record review after the participant gives birth. Participants randomized to the intervention arm will be provided with a fitbit, a sit-stand desk attachment, and will complete virtual health coaching visits every two weeks throughout pregnancy to facilitate reduced SED, increase standing, and increased stepping throughout the day.

ELIGIBILITY:
Inclusion Criteria:

* <13 w 0 d pregnant
* at risk for high levels of sedentary behavior: i) work at a desk job ≥ 30 hrs per week; ii) work at a desk job <30 hrs per week and report sitting on non-work days 1/2 the time or more; iii) do not work but report sitting 3/4 of the time or more; iv) self-reports <6000 steps per day
* ≥1 risk factor for APO: nulliparity, history of APO, prepregnancy BMI ≥ 30 kg/m2, or age ≥35 yr
* plan to deliver at UPMC facility or willing to provide medical record release for prenatal care and birth records

Exclusion Criteria:

* chronic hypertension (resting blood pressure ≥140/90 mmHg or antihypertensive medication use)
* pre-gestational diabetes
* self-report of inability to walk 2 blocks or climb a flight of stairs
* other serious medical condition in pregnancy for which exercise is contraindicated (e.g., underlying cardiac disease, severe anemia, chronic bronchitis, or poorly controlled hyperthyroidism or seizure disorder)
* unable to provide physician's consent to participate
* participating in another health-related intervention study that could affect study outcomes

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bethany B Gibbs, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Department of Health and Human Development, 32 Oak Hill Court, Room 220, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
The investigators do not have plans to share data at this time and will not be collecting biospecimens as part of this protocol. In the future, reasonable requests for de-identified data from other scientists will be considered. Such data will be shared with approval by the Study PI and other investigators, as appropriate.

REFERENCES:
- [Derived] Gibbs BB, Kozai AC, McAdoo SN, Davis KD, Savidge MB, Paley JL, Hauspurg A, Catov JM. The sedentary behavior reduction in pregnancy intervention (SPRING) pilot and feasibility randomized trial. BMC Pregnancy Childbirth. 2024 Apr 11;24(1):261. doi: 10.1186/s12884-024-06474-3. PMID 38605328
- [Derived] Barone Gibbs B, Kozai AC, McAdoo SN, Bastyr MC, Davis KD, Hauspurg A, Catov JM. Rationale, Design, and Methods for the Sedentary Behavior Reduction in Pregnancy Intervention (SPRING): Protocol for a Pilot and Feasibility Randomized Controlled Trial. JMIR Res Protoc. 2023 Jun 14;12:e48228. doi: 10.2196/48228. PMID 37314845

RESULTS

PARTICIPANT FLOW:
Recruitment Details: SPRING is a pilot and feasibility randomized clinical trial conducted in the greater Pittsburgh, PA (United States) area between October 2021 and June 2023.
Pre-assignment Details: A total of 51 first trimester pregnant individuals at risk for high sedentary behavior and adverse pregnancy outcomes (APO) were randomized 2:1 to a multi-component sedentary behavior reduction intervention or no-contact control.
Period: Overall Study
Arm/Group | Sedentary Behavior Reduction Intervention | Usual Care Control
Started | 34 (Randomized) | 17 (Randomized)
Completed | 27 (Completed 3rd trimester follow-up) | 15 (Completed 3rd trimester follow-up)
Not Completed | 7 | 2
Not completed — Pregnancy loss | 1 | 1
Not completed — Lost to Follow-up | 6 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sedentary Behavior Reduction Intervention | Usual Care Control | Total
Number analyzed (Participants) | 34 | 17 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (4.7) | 32.5 (3.6) | 32.1 (4.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 17 | 51
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 33 | 16 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 0 | 6
  White | 25 | 17 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Sedentary Time [Mean (Standard Deviation); unit: hours/day] — Total sedentary time spent in a 24-hour day
  hours/day | 10.42 (0.28) | 10.52 (0.40) | 10.47 (0.34)

OUTCOME MEASURES:

1. Primary Outcome: Sedentary Time
Description: objectively measured using activPAL3 micro
Time Frame: Randomization to study completion, about 6 months
Population: Two participants were removed from this analysis due to miscarriage after randomization.
Measure: Mean (Standard Deviation); unit: total hours/day
Arm/Group | Sedentary Behavior Reduction Intervention | Usual Care Control
Number analyzed (Participants) | 33 | 16
total hours/day
  Baseline Sedentary Time | 10.42 (0.28) | 10.52 (0.40)
  Follow-Up Sedentary Time | 9.62 (0.29) | 10.38 (0.34)
Statistical Analysis 1: Comparison: Sedentary Behavior Reduction Intervention vs Usual Care Control; Test type: Superiority; p < 0.05, Mixed Models Analysis

2. Primary Outcome: Standing
Description: Objectively measured using activPAL3 micro
Time Frame: Randomization to study completion, about 6 months
Population: Two participants were removed from this analysis due to miscarriage after randomization.
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Sedentary Behavior Reduction Intervention | Usual Care Control
Number analyzed (Participants) | 33 | 16
hours/day
  Baseline Standing | 2.79 (0.20) | 2.74 (0.29)
  Follow-Up Standing | 3.81 (0.26) | 2.81 (0.31)
Statistical Analysis 1: Comparison: Sedentary Behavior Reduction Intervention vs Usual Care Control; Test type: Superiority; p < 0.05, Mixed Models Analysis

3. Primary Outcome: Steps Per Day
Description: Objectively measured using activPAL3 micro
Time Frame: Randomization to study completion, about 6 months
Population: Two participants were removed from this analysis due to miscarriage after randomization.
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Sedentary Behavior Reduction Intervention | Usual Care Control
Number analyzed (Participants) | 33 | 16
steps per day
  Baseline Steps per day | 5224 (502) | 6268 (895)
  Follow-Up Steps per day | 6777 (656) | 6479 (919)
Statistical Analysis 1: Comparison: Sedentary Behavior Reduction Intervention vs Usual Care Control; Test type: Superiority; p < 0.05, Mixed Models Analysis

4. Secondary Outcome: Recruitment
Description: Participants screened for eligibility
Time Frame: Active recruitment phase, about 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Screened Candidates: Participants screened
Arm/Group | Screened Candidates
Number analyzed (Participants) | 140
Participants
  Pitt+Me Research Registry | 69
  Maternal Fetal Medicine Patient Referral | 38
  E-mail Advertisements to Pitt Community | 27
  Other (personal referrals, internet searches, and flyers) | 6
Statistical Analysis 1: Comparison: Screened Candidates; Test type: Other — Descriptive rates were calculated; Descriptive statistics only

5. Secondary Outcome: Retention
Description: Number of randomized intervention and control participants remaining at each follow up timepoint
Time Frame: Beginning of randomization to 2nd trimester and 3rd trimester
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Number of randomized intervention participants remaining in the trial at the third trimester study visit
- Control: Number of randomized control participants remaining in the trial at the third trimester study visit
Arm/Group | Intervention | Control
Number analyzed (Participants) | 34 | 17
Participants
  2nd Trimester Follow Up | 30 | 16
  3rd Trimester Follow Up | 27 | 15
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other — Descriptive statistics only; Descriptive statistics only

6. Secondary Outcome: Intervention Adherence to Behavioral Coaching Contacts
Description: Percentage of intervention contacts completed. This includes behavioral lessons and check-ins.
Time Frame: Randomization to study completion, about 6 months
Population: Initially, there were 34 Intervention participants. One participant was removed from this Intention To Treat analysis due to miscarriage after randomization.
Measure: Mean (Full Range); unit: percentage of contacts
Groups:
- Intervention: Multi-component sedentary behavior reduction
Arm/Group | Intervention
Number analyzed (Participants) | 33
percentage of contacts | 85.5 [70 to 94]
Statistical Analysis 1: Comparison: Intervention; Test type: Other — Descriptive statistics only; Descriptive statistics only

7. Secondary Outcome: Outcome Assessment Rates
Description: Number of participants that have complete objective sedentary time and other outcome data
Time Frame: Second and third trimester visit. Two participants were removed from this analysis due to miscarriage after randomization.
Population: Randomized participants with single gestation pregnancy
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Randomized to the behavioral intervention
- Control: Randomized to the control group
Arm/Group | Intervention | Control
Number analyzed (Participants) | 33 | 16
Participants
  2nd Trimester | 30 | 16
  3rd Trimester | 27 | 15
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other — Descriptive statistics only; Descriptive statistics only

ADVERSE EVENTS:
Time Frame: 3 Months
Description: Adverse events were collected from systematic questioning at assessment visits
Arm/Group | Sedentary Behavior Reduction Intervention | Usual Care Control
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/34 | 1/17
Other Adverse Events (participants affected / at risk) | 6/34 | 6/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sedentary Behavior Reduction Intervention (N=34) | Usual Care Control (N=17)
COVID (Infections and infestations) | 0 (0) | 1 (1) — Hospitalized due to headaches and increased liver enzymes
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sedentary Behavior Reduction Intervention (N=34) | Usual Care Control (N=17)
Mole Excision (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Benign mole excision from the bottom of foot
UTI (Infections and infestations) | 1 (1) | 0 (0) — Urinary Tract Infection
Neck, Spine, & TMJ Disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Prescribed physical therapy for neck, spine & TMJ pain related to past motor vehicle accident
Headaches & Nosebleeds (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Frequent headaches & nosebleeds
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1) — Increased heartburn concurrent with GI illness
Start of New Medication (Psychiatric disorders) | 0 (0) | 1 (1) — Began taking Zoloft for symptoms of irritability
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) — Food poisoning with emesis
Mild and general tailbone discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Symphysis Pubis Diastasis (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — Hospitalized and prescribed bedrest due to pubic symphysis joint separation
Sinus Infection (Infections and infestations) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) — Began treatment for depression
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) — Increased episodes of anxiety
Low Iron Level (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT05093842/Prot_SAP_000.pdf